CLINICAL TRIAL: NCT04528875
Title: Augmenting Ultrasound Imaging in Order to Replace Fluoroscopy in Image Guided Pain Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0266-19-RMB CTIL
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Image, Body
Keywords: ultrasound; imaging; lower back; CT, MRI
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound imaging — Imaging of low back with ultrasound

SUMMARY:
Utilizing existing data from CT/MRI images of patients, the investigators wish to develop an algorithm for augmenting the image obtained by ultrasound. In order to improved injection by ultrasound guidance

DETAILED DESCRIPTION:
Introduction:

A large proportion of injection-guided injections for pain relief including the lower back are performed with fluoroscopy. Performing the injection requires an adapted room, a fluoroscope with a C-shaped arm (c-arm), an X-ray technician, a physician, and a nurse. The amount of radiation, which is ionizing, is not negligible and depends very much on the reliability of the medical team. The injections performed in this technique include injections into the epidural space, injections into the facet joints (joints between the vertebrae of the back), nerve blocks, and radiofrequency nerve ablation.

Using ultrasound imaging, as a substitute for fluoroscopy, may help real-time guidance of needle placement, and allow imaging from multiple directions, without ionizing radiation that endangers the patient and caregivers, while reducing treatment. costs The use of ultrasound imaging will allow these treatments to be performed in outpatient clinics as well, without the need for expensive equipment.

Nowadays, with the existing ultrasound equipment, there is a very high variability as to the quality of the image obtained while scanning the lower back. Poor image quality makes it very difficult to perform an accurate and reliable injection. In contrast, the structures of the lower back can be optimally simulated using CT (mainly the skeletal structures such as vertebrae and joints) and using MRI (better resolution for soft tissue structures than for skeletal structures). Performing invasive injections under the guidance of these measures is costly both in terms of equipment and in terms of manpower and certainly contributes to ionizing exposure in the case of CT. At the same time, many patients come to the Institute of Pain Medicine, after performing these imaging tests.

The investigators intend to develop an algorithm in which these tests (CT, MRI) will serve as a database for each patient participating in the study whose back will be scanned using an ultrasound transducer. According to the initiators of the study, the investigators can develop an imaging application that will rely on both the information of an imaging image of CT and / or MRI and after the back scan (using an ultrasound transducer) the investigators will get an improved (augmented) ultrasound image that can be used in the future as an ultrasound-guided injection.

The aim of the present study is to improve the quality of the imaging image obtained when scanning the lower back with an ultrasound transducer using the information available from previous imaging images - CT and / or MRI

The study population:

Patients who are referred to the Rambam Institute of Pain Medicine suffering from low back pain and who have already undergone a CT scan or MRI examination of the lower back before arriving at the Institute

Number of participants in this center:

50 patients

Age range:

Between the ages of 18 and 80

Gender:

Without gender restriction

Criteria for inclusion:

1. Low back pain including lower / upper back pain.
2. Patients who underwent MRI or CT imaging of the lower back during the past year.
3. Patients who can understand the rationale of the study and can sign an informed consent form.

Criteria for exclusion:

1. Back surgery in the lower back area
2. Significant deformity in the back such as scoliosis with an angle above 50 degrees

Criteria for removal from the experiment:

none

The duration of the medical trial includes the follow-up period after the trial:

About a year

Clinical follow-up program (during and after treatment):

A: Patients eligible for the study will receive an explanation and sign a scientific consent form.

B: Subjects will fill out a short demographic questionnaire as well as a questionnaire about their pain problem. Each subject will receive a unique identification number for the study itself.

C: The subjects will be admitted to the Institute of Pain Medicine for the purpose of scanning the back using an ultrasound device. The required imaging acquisition, using the standard transducer (curved array or phased array), is of three scans along the bilateral spine, and three transverse scans in the same area. After scanning - which will take about 5 minutes, the data will be stored in digital media anonymously but with the unique identification number given to the patient in section B.

D: The digital media - CT or MRI will be uploaded to the hospital's imaging archive. Data will be transferred anonymously to external media (disk with a unique identification number of the study only) The digital information of both the ultrasound scan and the previous imaging tests will be transferred to a biotechnology lab, without any identifying details of the patient for analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients with low back pain including lower / upper back pain. Patients who underwent MRI or CT imaging of the lower back during the past year.

Patients who can understand the rationale of the study and can sign an informed consent form.

Exclusion Criteria:

Patients who have undergone back surgery in the lower back area Patients with significant deformity (deformity) in the back such as scoliosis with an angle above 50 degrees

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are referred to the Rambam Institute of Pain Medicine suffering from low back pain and who have already undergone a CT scan or MRI examination of the lower back before arriving at the Institute
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Algorithm for imaging augmentation of ultrasound | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon Vulfsons, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No